CLINICAL TRIAL: NCT05829902
Title: Evaluation of an Herbal Extract on Sleep Parameters in Healthy, Middle-aged Women
Brief Title: Evaluation of an Herbal Extract on Sleep Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aventure AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sleepwell_2023
Record Dates: First submitted 2023-03-29; First posted 2023-04-26 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Sleep Onset Latency
Keywords: Sleep Onset Latency (SOL); Herbal extract; Lemon balm

STUDY DESIGN:
Intervention Model Description: This study is a randomized, placebo-controlled, parallel intervention with two arms. The study is divided into three phases: the run-in period (14 days), the intervention period (14 days) and the follow-up period (14 days). Eligible participants will be randomized in a 1:1 ratio to receive either lemon balm extract or a placebo. Randomization will be stratified by ISI-value and age at baseline. Treatment assignments will be pre-planned according to a computer-generated randomization scheme prepared by a vendor.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A copy of the randomization list will be provided to those packing the product kits. The randomization list is a document that consists of randomization numbers, which uniquely assign each study patient to one of the treatments. The sponsor and all staff directly involved in the trial will thus be blinded to the product allocated to the participants. The randomization number will be documented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active product (Experimental): The active product is a drink consisting of 600 mg of lemon balm extract, tea leaves, brown sugar and powdered flavoring agent that is mixed with lukewarm water. The volume per serving is 30 ml. The drink will be taken every night before sleep for a period of two weeks.
  Interventions: Other: Herbal extract drink
- Placebo (Placebo Comparator): The placebo drink is maltodextrin mixed with water, and the same tea leaves, brown sugar and powdered flavoring agent as the test drink. The volume per serving is 30 ml. The drink will be taken every night before sleep for a period of two weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Herbal extract drink — 30 ml drink containing 600 mg of lemon balm extract, tea leaves, brown sugar and flavoring agent, two weeks daily
  Arms: Active product
Other: Placebo — 30 ml placebo drink containing maltodextrin, tea leaves, brown sugar and flavoring agent, two weeks daily
  Arms: Placebo

SUMMARY:
The overall purpose of this interventional study is to investigate how a specific herbal extract influences the quality of sleep in middle-aged women with mild to moderate insomnia. During the study, the participants are asked to take the test drink every night for two weeks. Both objective (Oura ring) and subjective (analog sleep diaries, questionnaires) measures are included to evaluate sleep parameters as well as perceived alertness and impact on daily functions. The primary outcome is sleep onset latency (SOL), which is the time it takes for a person to fall asleep. Secondary outcomes which will be evaluated include time spent in different sleep stages, number of times waking up during the night, and various qualitative ratings of energy levels and mood during the day.

Researchers will compare the group with active product and placebo product to see if the consumption of the herbal extract will lead to improvements in the factors mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 35-60
* BMI 18-30 kg/m2
* Mild to moderate insomnia according to the ISI (Insomnia Severity Index) questionnaire (ISI-value 10-21)
* Matching results from the Oura ring and sleep diaries during the run-in period

Exclusion Criteria:

* Metabolic disease (diabetes, cardiovascular disorders, hypo- or hyperthyroidism, etc)
* Severe psychiatric disorders
* Pregnancy, breastfeeding
* Restless legs or leg cramps that influence sleep and everyday life
* Conditions that prevent sleep through the symptoms that they produce (pain, nightly coughs, etc)
* Breathing problems (asthma, severe snoring, sleep apnea, etc)
* Medication that can influence sleep and/or wakefulness
* Consumption of herbal sedatives during the last month
* Having someone in the household that needs to be tended to during the night and pose a major risk to disturb the research participant's sleep to a large extent.
* Irregular work hours, including shift work at night
* Regularly sleeping more than 1 night per week away from home
* Tobacco or drug use
* Other factors that are deemed to influence participation negatively

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Sleep onset latency | 2 weeks
  The length of time it takes a person to fall asleep when turning the lights off, this parameter will be measured by using the Oura Ring

SECONDARY OUTCOMES:
Time spent in different sleep stages | 2 weeks
  These Parameters will be measured by using the Oura Ring
Perceived alertness and wellbeing during the day | 2 weeks
  These parameters will be measured by using a sleep diary (pen and paper) with a ranking scale which needs to be filled out in the morning and in the evening

CONTACTS AND LOCATIONS:
Locations (1):
- Aventure Clinical Trial Unit, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No